CLINICAL TRIAL: NCT01238809
Title: Gastroprotective Agent Utilization and Compliance in Patients > 60 Years Taking Low-dose Aspirin in France
Status: Withdrawn | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CFR-DUM-2010/1
Record Dates: First submitted 2010-11-09; First posted 2010-11-11 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Self-administered Questionnaire to Patients
Keywords: Compliance; France
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to assess in general population low-dose aspirin and gastroprotective agent compliance and reasons for bad compliance

ELIGIBILITY:
Inclusion Criteria:

* French people > 60 years old, part of Kantar Health Access Sant� panel

Exclusion Criteria: -

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 7300 (Estimated)
Dates: Start 2011-06; Primary Completion 2011-07 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
low-dose aspirin and gastroprotective treatment compliance (Girerd questionnaire: a 6-item self-administered and validated questionnaire to evaluate adherence to treatments) | One month

CONTACTS AND LOCATIONS:
Overall Officials: Mrs Genevieve BONNELYE, Principal Investigator — KantarHealth - France